CLINICAL TRIAL: NCT05506774
Title: A Multi-centre, Non-interventional Retrospective Study to Describe Treatment Pathways, Outcomes, and Resource Use in Patients With CD30 Positive Lymphoma in China (REALM)
Brief Title: A Study of People With CD30 Positive Lymphoma in China
Acronym: REALM
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C25028
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Lymphoma
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Participants With cHL.: Participants who diagnosed with cHL between January 1, 2018 and March 31, 2021, and have demographic and clinical data available in hospital information system (HIS)/electronic medical records (EMRs) or laboratory information management will be observed retrospectively from the date of diagnosis with cHL until death, loss to follow-up, or end of the study, whichever occurs first.
- Cohort B: Participants With NHL.: Participants who diagnosed with NHL between January 1, 2018 and March 31, 2021, and have demographic and clinical data available in HIS/EMRs or laboratory information management will be observed retrospectively from the date of diagnosis with NHL until death, loss to follow-up, or end of the study, whichever occurs first.

SUMMARY:
The main aim is to see how adult participants with newly diagnosed or relapsed/refractory CD30+ lymphoma responded to any previous treatment in China.

The study sponsor will not be involved in how participants are treated, the study only consists of collecting demographic and clinical records information from the hospital clinical systems. Based on the diagnosis of the disease, participants will be assigned to one of the following groups and their information will be analyzed within that group respectively:

* Group A: Participants diagnosed with classical Hodgkin lymphoma (cHL).
* Group B: participants diagnosed with non-Hodgkin lymphoma (NHL), including systemic anaplastic large-cell lymphoma [sALCL], peripheral T-cell lymphoma-not otherwise specified [PTCL-NOS], angioimmunoblastic T-cell lymphoma [AITL], extranodal NK/T-cell lymphoma [ENKTCL], mycosis fungoides [MF], primary cutaneous anaplastic large cell lymphoma [pcALCL], diffuse large B-cell lymphoma [DLBCL], primary mediastinal B-cell lymphoma [PMBCL]).

DETAILED DESCRIPTION:
This is an observational, non-interventional, retrospective study in participants with newly diagnosed or relapsed/refractory CD30+ lymphoma to describe the treatment pathways, outcomes, and resource use among adult participants.

The study will enroll approximately 2800 participants. The data will be collected from participants' medical records between January 1, 2018 and March 31, 2021 and recorded in the in case report forms (CRFs). Participants will be assigned to the following two observational cohorts based on pathological diagnosis:

* Cohort A: Participants with cHL
* Cohort B: Participants with NHL

This multi-center trial will be conducted in China. All participants will be observed for at least 6 months or until death, loss to follow-up, or end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion criteria:

1. Who newly diagnosed with or refractory/relapsed with cHL, sALCL, CD30+ non-sALCL-NHL confirmed by immunochemistry with any CD30 expression (that is, PTCL-NOS, AITL, ENKTCL, MF, pcALCL, DLBCL, PMBCL) between January 1, 2018 and March 31, 2021 and only one CD30+ pathology report will be needed for CD30+ non-sALCL-NHL.
2. Who have received anti-lymphoma treatment between January 1, 2018 and March 31, 2021.

Exclusion criteria:

1. Whose demographics and clinical features are not available from medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with CD30+ lymphoma (newly diagnosed or refractory/relapsed) and treated between January 1, 2018 and March 31, 2021 will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1006 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Different Initial Treatments Based on Different Lines of Therapy | At Day 1 of initial treatment
  The initial treatment is defined as the first treatment information after enrolment during the data collection, regardless of treatment lines. Initial treatments will include but not limited to the following: chemotherapy, radiotherapy, targeted therapy, immunotherapy, autologous stem cell transplant (ASCT), and other treatments). Different lines of therapy will include the following: the initial treatment in first-line (newly diagnosed), second-line (first refractory/relapsed), and third- or later-line (refractory/relapsed after 2 or more lines of therapies).

SECONDARY OUTCOMES:
Number of Participants Categorized Based on Clinical Characteristics | Up to 2 months before the index date
  Index date is defined the first treatment initiation date after enrollment regardless of treatment lines. The initial treatment is defined as the first treatment information after enrolment during the data collection, regardless of treatment lines. Clinical characteristics include the clinical staging of adult participants with initial diagnosis or relapsed/refractory CD30+ lymphoma in China will be reported.
Real World Overall Response Rate (rwORR) | Up to 3 years and 9 months
  The rwORR is defined as the percentage of participants who achieve complete response (CR) or partial response (PR) assessed by clinician documented in EMRs after the initial treatment. The rwORR will be determined by positron emission tomography-computed tomography (PET-CT) and computed tomography (CT) based on response criteria as per Lugano 2014.
Real World Progression Free Survival (rwPFS) | Up to 3 years and 9 months
  rwPFS is defined as the time from the initial treatment to the documented of relapsed or disease progression or death due to any cause, whichever occurs first. It will be analyzed using Kaplan-Meier method. The rwPFS will be determined by PET-CT and CT based on response criteria as per Lugano 2014.
Real World Overall Survival (rwOS) | Up to 3 years and 9 months
  rwOS is defined as the time from the date of initial treatment to the date of death from any cause. It will be analyzed using Kaplan-Meier method.
Duration of Hospital Stay Based on Different Lines of Therapy | Up to 3 years and 9 months
  Different lines of therapy will include the following: the initial treatment in first-line (newly diagnosed), second-line (first refractory/relapsed), and third- or later-line (refractory/relapsed after 2 or more lines of therapies). The duration of hospital admission will be reported and categorized based on different lines of therapy.
Number of Hospitalization Based on Different Lines of Therapy | Up to 3 years and 9 months
  Different lines of therapy will include the following: the initial treatment in first-line (newly diagnosed), second-line (first refractory/relapsed), and third- or later-line (refractory/relapsed after 2 or more lines of therapies). The number of hospital admission will be reported and categorized based on different lines of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- China (11):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Union Hospital AffiliatedProf to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital/the Firstaffiliated Hospital Withnanjing Medical University, Nanjing, Jiangsu
  - The Firstaffiliated Hospital Ofsoochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Provincial Hospital Affiliated to Shandong First Medical University (Shandong Provincial Hospital), Shandong, Jinan
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/